CLINICAL TRIAL: NCT04248699
Title: Open-Label Study to Assess the Impact of Lycored's Nutritional Supplement Lumenato on Skin Parameters in Healthy Women
Brief Title: Lumenato Nutritional Supplement on Skin Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Collaborators: ObvioHealth (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBVIO-LYC-002
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-01

CONDITIONS: Skin
Keywords: Nutritional Supplement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumenato Supplement (Experimental): tomato oleoresin
  Interventions: Dietary Supplement: Lumenato

INTERVENTIONS:
Dietary Supplement: Lumenato — tomato oleoresin obtained from yellow dry tomato pulp

SUMMARY:
This 12-week study is an open-label study assessing the perceived effectiveness of the Lycored Lumenato supplement on skin health and appearance.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate perceived changes in skin health and appearance after taking the study product daily for 12 weeks. The study product is a soft gel supplement containing tomato oil. This an open-label study, meaning there is no placebo control arm for the study, and everyone enrolled in the study will receive the active study product.

ELIGIBILITY:
Inclusion criteria:

* Resides in the United States
* Generally healthy women between the ages of 35-55
* Fitzpatrick skin types 2 or 3
* Identifies as one of the following: Asian, White, Hispanic/Latino, or both White and Hispanic/Latino
* Type 2 on the Glogau Skin Classification scale
* Has expressed interest in improving skin health and appearance
* Willing and able to follow the procedures of the study
* Willing to refrain from changing their diet or lifestyle significantly for the duration of the study
* Able to understand the study requirements and activities in English, and provide informed consent
* Access to reliable internet service and smartphone in order to utilize the ClaimIt software/app needed to remotely participate in the study

Exclusion Criteria:

* Participants with Fitzpatrick skin types of 1, 4, 5 or 6
* Known allergies or sensitivity to tomato, latex and/or potato
* Current use or use within 1 month of study enrollment of hormonal therapies (including hormonal contraceptives)
* Current, regular use or regular use within 1 month of study enrollment of oral steroids; regular use defined as >10 consecutive days
* Chronic or relapsing inflammatory and/or allergic skin conditions such as atopic dermatitis, rosacea, psoriasis and alike including telangiectasias ("spider veins")
* Pregnant, lactating or breastfeeding women (within the last 6 months) or those planning to become pregnant during the study period
* Less than 2 years since diagnosis or treatment of skin cancer including basal cell carcinoma, squamous cell carcinoma, melanoma- excluding actinic keratosis
* Currently active herpes infections or currently on treatment for herpes infections
* History of facial keloids
* Current diagnosis of adult acne or currently on treatment for adult acne
* Recent (<6 months at enrollment) cardiovascular conditions such as stroke, transient ischemic attack (TIA), or myocardial ischemia/infarction, recently on treatment for congestive heart failure, or currently having vasculitis or vascular conditions
* On potent blood thinners such as low-molecular weight heparin (LMWH), rivaroxaban, apixaban, or other prescription blood thinners - excludes aspirin
* Holds a current diagnosis of diabetes mellitus type I or II
* Participants who have received facial irradiation within last year or are planning on undergoing facial irradiation during the study
* Chronic liver disease- excluding early stage non-alcoholic fatty liver disease (NAFLD)
* Chronic kidney disease or recent (<6 months at enrollment) acute kidney disease
* Participants who currently take supplements containing carotenoids, lutein, melatonin or tryptophan
* Participants with occupations or lifestyle that require significant daily exposure to the sun (defined as at least 1 hour of continuous outdoor sun exposure)
* Participants who have had a sunburn in the last 2 weeks
* Participants who use tanning salons or tanning products in the last 3 months
* Participants who plan to undergo invasive facial procedures (injections, chemical peeling, etc.) during the study or have undergone these procedures within 2 months prior to enrollment
* Change in oral supplements or medications targeting skin health within 2 months prior to enrollment
* Participants who are HIV positive
* Participants who are immunosuppressed
* Participants with a recent (<2 months prior to enrollment) diagnosis of a psychiatric condition
* Participants having chronic connective tissue disorder affecting the skin (e.g. Ehlers- Danlos syndrome, Marfan's Syndrome, Osteogenesis Imperfecta)
* Participants with auto-immune skin diseases (e.g. scleroderma, psoriasis, lupus, epidermolysis bullosa, bullous pemphigoid, temporal arteritis)
* Participants who have been prescribed retinoids treatment (<2 months prior to enrollment)
* Participants who meet either/or both of the following criteria with regards to smoking habits (smoking includes cigarettes, e-cigs, pipes, hookah, cigars):
* Who are current smokers (smoked at least 100 cigarettes, or tobacco/nicotine equivalent, in her lifetime) and who continue to use these products
* Who were former smokers (smoked at least 100 cigarettes, or tobacco/nicotine equivalent, in her lifetime, but who have quit smoking) who have smoked within the last year and/or were former smokers for 10 years
* Participants who drink more than 14 drinks per week (more than 2 drinks per night)
* Participants who use illicit or illegal drugs
* Participants who are regular users of cannabis substances or substances derived from cannabis such as CBD, CBD oils or balms, cannabis-containing edibles; vaping; smoking; hookahs.
* NOTE: regular use is defined as long stretches of inhaling or consuming these products over several months or longer. Occasional, but not weekly, use of products with small amounts of CBD-related compounds (e.g. waters with CBD infusions) are not considered regular use.)
* Participants who are planning a trip to the mountains or to a higher UV index region during the study period
* Any other medication, condition or disease that in the PI's opinion that may adversely affect the participant's ability to complete the study, substantially impact the study's integrity or may pose a significant risk to the participant
* Participants who are experiencing perimenopausal or menopausal symptoms
* Participants who have had a hysterectomy and/or both of their ovaries removed

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Participant perception of the improvement in skin health and appearance from Baseline to Week 12 using the questionnaire responses from FACE-Q™ | 12 weeks
  FACE-Q™ Satisfaction with Skin scale: gathers the participant perspective of their satisfaction or dissatisfaction with their facial skin using a 12-question scale. Participants are asked to choose one of the following responses for each question: Very Dissatisfied (1), Somewhat Dissatisfied (2), Somewhat Satisfied (3) and Very Satisfied (4) for each 12 questions and the sum of scores (or mean of the completed items, in the event of an incomplete scale) gets converted into a score from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Baseline Skin Questionnaire | 12 weeks
  Participant perception of change or maintenance in a variety of skin health parameters over the course of the study using the subjective "Baseline Skin Questionnaire"
End of Study Product Questionnaire" | 12 weeks
  Participant perception of the study product and study experience as assessed by the "End of Study Product Questionnaire"
Skin Update Questionnaire | 12 weeks
  Participant perception of change or maintenance in a variety of skin health parameters over the course of the study using the subjective "Update Skin Questionnaire"

OTHER OUTCOMES:
Adverse events (AEs) observed during the study, classified by the investigator as to severity, relationship to the study product/protocol, and seriousness | 14 weeks
  classified by the investigator
Compliance to the daily use of the Lycored Lumenato supplement through monitoring within ClaimIt (Weekly e-Diary) | 12 weeks
  Weekly e-Diary
Sustainability of effect after two weeks without supplementation as assessed by the Week 14 FACE-Q™ Satisfaction with Skin scale | 14 weeks
  FACE-Q™ Satisfaction with Skin scale: gathers the participant perspective of their satisfaction or dissatisfaction with their facial skin using a 12-question scale. Participants are asked to choose one of the following responses for each question: Very Dissatisfied (1), Somewhat Dissatisfied (2), Somewhat Satisfied (3) and Very Satisfied (4) for each 12 questions and the sum of scores (or mean of the completed items, in the event of an incomplete scale) gets converted into a score from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, MD, Principal Investigator — ObvioHealth
Locations (1):
- o ObvioHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glogau RG. Aesthetic and anatomic analysis of the aging skin. Semin Cutan Med Surg. 1996 Sep;15(3):134-8. doi: 10.1016/s1085-5629(96)80003-4. PMID 8948530
- [Background] Groten K, Marini A, Grether-Beck S, Jaenicke T, Ibbotson SH, Moseley H, Ferguson J, Krutmann J. Tomato Phytonutrients Balance UV Response: Results from a Double-Blind, Randomized, Placebo-Controlled Study. Skin Pharmacol Physiol. 2019;32(2):101-108. doi: 10.1159/000497104. Epub 2019 Mar 5. PMID 30836363
- [Background] Havas F, Krispin S, Melendez-Martinez AJ, von Oppen-Bezalel L. Preliminary Data on the Safety of Phytoene- and Phytofluene-Rich Products for Human Use including Topical Application. J Toxicol. 2018 Apr 15;2018:5475784. doi: 10.1155/2018/5475784. eCollection 2018. PMID 29849613
- [Result] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516